CLINICAL TRIAL: NCT05799456
Title: Glycosaminoglycan Scores as Early Detection Biomarkers in Bladder Urothelial Carcinoma
Status: Completed | Type: Observational
Sponsor: Jens Nielsen (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor-Investigator, Jens Nielsen, Professor, Chalmers University of Technology
Organization: Chalmers University of Technology (Other)
Other Study IDs: GAG-BCa-001
Record Dates: First submitted 2023-03-20; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bladder cancer
  Interventions: Diagnostic Test: Free glycosaminoglycan profiling
- No evidence of disease
  Interventions: Diagnostic Test: Free glycosaminoglycan profiling

INTERVENTIONS:
Diagnostic Test: Free glycosaminoglycan profiling — Free glycosaminoglycan profiling (GAGome) analysis was performed at a single blinded central laboratory using commercial kits wherein the concentration (in µg/mL) of 17 chondroitin sulfate (CS), heparan sulfate (HS), hyaluronic acid (HA) disaccharides were detected and quantified using a UHPLC-MS/MS system.

SUMMARY:
Early detection of bladder cancer (BCa) is considered an effective strategy to curb mortality from the disease. However, current urinary biomarkers have insufficient specificity to warrant BCa screening. Urine free glycosaminoglycan profiles (or GAGomes) are promising noninvasive biomarkers of cancer metabolism. In this study, samples are obtained from patients with BCa and controls to compare the glycosaminoglycan profiles between groups.

ELIGIBILITY:
Cases (Bladder cancer [BCa])

Inclusion Criteria:

* Primary BCa diagnosis at cystoscopy, planned for TURB

Exclusion Criteria:

* No histopathological diagnosis of BCaTa-T4 N0-2 MX-0 after TURB

Controls (No evidence of disease [NED])

Inclusion Criteria:

* In follow-up with cystoscopy after treatment Ta-T3 N0-2 M0 BCa or upper tract urothelial cancer no evidence of disease at cystoscopy for at least 6 months prior to inclusion
* No history of cancer except urothelial

Exclusion Criteria:

* Positive cytology at inclusion visit
* Intravesical instillation therapy during 6 months prior to inclusion visit

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective case-control study to compare patients elected for transurethral resection of the bladder (TURB) for bladder cancer (BCa) [cases] versus patients with no evidence of disease (NED) during the follow-up of previously localised BCa [controls].
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Area-under-the-receiving operating characteristic (ROC)-curve (AUC) for the classification of BCa versus NED | Before primary surgery for BCa; at a post-surgical follow-up visit for controls up to 5 years from primary surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Institute of Clinical Science, Sahlgrenska Academy, University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No